CLINICAL TRIAL: NCT04589312
Title: The Safety and imMunogeNicity of Combined Pertussis-cOntaining Vaccine (Tdap) for HIV-infected Pregnant WomEn and Their newboRns - A Randomized Clinical Trial
Brief Title: Maternal Pertussis Wholecell Responses
Acronym: WoMANPOWER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: Medical Research Council (Other Government); University of British Columbia (Other); Public Health England (Other Government); MU-JHU CARE (Other); BioNet-Asia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17.0019
Record Dates: First submitted 2020-10-01; First posted 2020-10-19 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pertussis
Keywords: Whooping Cough; Pertussis; Vaccination; Pregnancy; Infant; Newborn; HIV
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Intervention Model Description: The study will take a 2x2 formation, with four groups:
  1. HIV-uninfected women, standard of care vaccines in pregnancy;
  2. HIV-uninfected women, Tdap vaccine in pregnancy;
  3. HIV-infected women, standard of care vaccines in pregnancy;
  4. HIV-infected women, Tdap vaccine in pregnancy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study nursing staff and participants will be blinded to the vaccine given and vaccine syringes will be covered with an opaque label, obscuring the vaccine. Only the preparing pharmacist will be aware of the vaccine used. A study nurse who is blinded to the vaccine given will observe for immediate reactions to the vaccine in a separate room from where the woman will receive her vaccination. This room will have an emergency trolley with appropriate drugs available should these be required.
  The laboratory-based research team conducting the assays will be blinded to subject allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pregnant women not living with HIV, Td vaccine (Active Comparator)
  Interventions: Biological: Standard of care vaccines
- Pregnant women not living with HIV, Tdap vaccine (Experimental)
  Interventions: Biological: Boostagen, (BioNet-Asia)
- Pregnant women living with HIV, Td vaccine (Active Comparator)
  Interventions: Biological: Standard of care vaccines
- Pregnant women living with HIV, Tdap vaccine (Experimental)
  Interventions: Biological: Boostagen, (BioNet-Asia)

INTERVENTIONS:
Biological: Standard of care vaccines — Visit 1: Check tetanus immunisation status. Vaccination up to 25+ 6 weeks of pregnancy with Td; Visit 2: vaccination at least 4 weeks after visit 2 with either Tdap or Td (per randomisation and according to WHO guidance)
  Arms: Pregnant women living with HIV, Td vaccine; Pregnant women not living with HIV, Td vaccine
Biological: Boostagen, (BioNet-Asia) — Visit 1: Check tetanus immunisation status. Vaccination up to 25+ 6 weeks of pregnancy with Td; Visit 2: vaccination at least 4 weeks after visit 2 with either Tdap or Td (per randomisation and according to WHO guidance);
  Arms: Pregnant women living with HIV, Tdap vaccine; Pregnant women not living with HIV, Tdap vaccine

SUMMARY:
Pertussis is resurging worldwide. In Africa alone it is estimated that there are 2.1 million cases and 542,000 deaths from pertussis in infants under 1 year with the highest rates of morbidity and mortality in infants <3 months old, before possible prevention via the infant immunization programme1. To protect these most vulnerable infants, the World Health Organisation (WHO) recommends Tdap vaccination as safe in pregnancy and recommends the use of wP vaccines within the EPI. Maternal antibody following aP vaccination can interfere with infant anti-pertussis antibody responses post infant EPI vaccination, which is of concern in high burden settings such as Uganda. There are therefore multiple factors in this population which may influence the effect of pertussis immunization in pregnancy, and which have not been studied, most notably HIV infection and interference with wP vaccines in infants. The immunogenicity of Tdap in HIV-infected pregnant women has not yet been examined. In addition, to date, the effect of maternal vaccination, placental transfer and infant antibody responses in HEU infants have not been studied at all. There are no studies examining the immune response to wP vaccine administered to infants (EPI recommendation) whose mothers received aP in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a woman aged 18 years or older, inclusive at day of signing the ICF;
* Pregnant woman at >16 and <26 weeks gestation, verified by ultrasound scan;
* Documented HIV test during pregnancy taken by rapid test at the screening visit;
* Low risk, singleton pregnancy, as assessed by the study physician based on ultrasound scan and previous obstetric history; and
* The woman is willing to comply with the study procedures, including giving birth at Kawempe National Referral Hospital, remaining in the study area until the infant is 1 year old and is able to provide informed consent for herself and on behalf of the infant

Exclusion Criteria:

Any of the following:

* Previous anaphylaxis to any component of Td or Tdap vaccines;
* vaccination is otherwise contraindicated (per product monographs);
* Documented to have received four or more previous tetanus toxoid vaccine doses (as this would prevent randomisation to Tdap group and receipt of two additional tetanus toxoid containing vaccines);
* History of pre-eclampsia or eclampsia in previous pregnancies;
* Gestational diabetes in current pregnancy;
* Rhesus negative mothers;
* Multigravida;
* Previous late stillbirth (defined as loss of pregnancy at any time after 28 weeks gestation);
* Previous low birth weight baby of less than 2.0 kilograms or premature delivery (defined as a delivery before 37 weeks gestation);
* Previous neonatal death (defined as death of an infant within the first 28 days of life);
* Previous delivery of an infant with a known or suspected genetic or chromosomal abnormality;
* History of other significant pregnancy related complications judged likely to affect the safety of the mother or infant or to significantly compromise the endpoint data collected;
* History of other significant neonatal complications judged likely to affect the safety of the mother or infant or to significantly compromise the endpoint data collected;
* Significant maternal chronic illness including but not limited to hypertension requiring treatment, heart disease, lung disease, neurological disorders including a history of epilepsy or recurrent afebrile seizures, kidney disease, liver disease, anaemia and other haematological disorders (including sickle cell), endocrine disorders including known diabetes mellitus, autoimmunity;
* Severe anaemia (less than 7.0g/dL);
* Known Syphilis or hepatitis B (HBV) virus positive or found to be Syphilis or HBV positive during screening;
* Any other condition judged to significantly increase the risks to either the mother or the infant within the current pregnancy (including relevant history from previous pregnancies);
* Receipt of any blood product including human immunoglobulins at any stage during the current pregnancy or plan to receive any blood products during the period or trial participation (receipt of blood products in an emergency or for obstetric reasons will not represent a protocol deviation given such situations are unplanned);
* Clinically suspected or confirmed congenital or acquired clotting or bleeding disorders or the current receipt of medications known to alter clotting or bleeding;
* Any clinically significant signs or symptoms of acute illness, significant abnormalities in vital signs, an axillary temperature of greater than 38.0°C or any recorded fever (greater than 38.0°C) in the preceding 24 hours;
* Two or more symptoms (nausea/vomiting, diarrhoea, headaches, fatigue and myalgia) rated as grade 2 and clinically significant on the maternal systemic reactogenicity scale present at baseline on the day of vaccination;
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily;
* Participation in the 4 weeks preceding the trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure;
* History of being treated for pertussis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Anti-pertussis toxin (PT) and anti-FHA IgG concentrations in cord blood of Tdap-vaccinated HIV-infected vs HIV-uninfected pregnant women. | At delivery
Anti-pertussis toxin (PT) and anti-FHA IgG concentrations in cord blood of Tdap -vaccinated vs Tdap -unvaccinated pregnant women and whether this differs by maternal HIV status. | At delivery
Anti-PT and anti-FHA IgG concentrations in infants born to Tdap vaccinated vs Tdap -unvaccinated pregnant women 4 weeks after the completion of a series of primary vaccination with 3 doses of wP vaccine, and whether this differs by maternal HIV status. | 18 weeks of pregnancy
Safety Outcome: Safety assessment of Tdap vaccine vs Td vaccine in HIV-infected vs HIV-uninfected pregnant women - Pregnant Women | First vaccination visits
  Percentage of maternal Subjects With Solicited Local and Solicited Systemic AEs and percentage with any Unsolocited AEs; Percentage of Maternal Subjects With Serious Adverse Events (SAEs), Unsolicited Medically Attended AEs (MAEs) and Unsolicited AEs Leading to Study Withdrawal
Safety Outcome: Safety assessment of Tdap vaccine vs Td vaccine in HIV-infected vs HIV-uninfected pregnant women - Pregnant Women | At 12 months of age of infants
  Percentage of maternal Subjects With Solicited Local and Solicited Systemic AEs and percentage with any Unsolocited AEs; Percentage of Maternal Subjects With Serious Adverse Events (SAEs), Unsolicited Medically Attended AEs (MAEs) and Unsolicited AEs Leading to Study Withdrawal
Safety Outcome: Safety assessment of Tdap vaccine vs Td vaccine in HIV-infected vs HIV-uninfected pregnant women - Infants | At birth
  Percentage of Infants With SAEs, Unsolicited AEs and AEs Leading to Study Withdrawal by a clinical examination
Safety Outcome: Safety assessment of Tdap vaccine vs Td vaccine in HIV-infected vs HIV-uninfected pregnant women - Infants | At 18 weeks of age
  Percentage of Infants With SAEs, Unsolicited AEs and AEs Leading to Study Withdrawal by a clinical examination
Safety Outcome: Safety assessment of Tdap vaccine vs Td vaccine in HIV-infected vs HIV-uninfected pregnant women - Infants | At 6 months of age to assess health of the infant (phone call)
  Percentage of Infants With SAEs, Unsolicited AEs and AEs Leading to Study Withdrawal by a clinical examination
Safety Outcome: Safety assessment of Tdap vaccine vs Td vaccine in HIV-infected vs HIV-uninfected pregnant women - Infants | At 9 months of age to assess health of the infant (phone call)
  Percentage of Infants With SAEs, Unsolicited AEs and AEs Leading to Study Withdrawal by a clinical examination
Safety Outcome: Safety assessment of Tdap vaccine vs Td vaccine in HIV-infected vs HIV-uninfected pregnant women - Infants | At 12 months of age to assess health of the infant (phone call)
  Percentage of Infants With SAEs, Unsolicited AEs and AEs Leading to Study Withdrawal by a clinical examination

SECONDARY OUTCOMES:
Anti-PT and anti-FHA IgG concentrations in HIV-infected and HIV-uninfected pregnant women following Tdap vs Td vaccination during pregnancy (4 weeks post-vaccine & at delivery) | 4 weeks post-vaccine & at delivery
Anti-PT IgG antibody avidity in HIV-infected and HIV-uninfected pregnant women following Tdap vs Td vaccination during pregnancy | 18 weeks of pregnancy, 4 weeks post-vaccine, at delivery
Serum bactericidal activity in HIV-infected and HIV-uninfected pregnant women following Tdap vs Td vaccination during pregnancy | 18 weeks of pregnancy, 4 weeks post-vaccine, at delivery
Anti-PT IgG and anti-FHA placental transfer ratios in HIV-infected and HIV-uninfected pregnant women following Tdap vs Td vaccination during pregnancy | 18 weeks of pregnancy, 4 weeks post-vaccine, at delivery
Tetanus Toxoid antibody responses in HIV-infected and HIV-uninfected pregnant women following Tdap vs Td vaccination during pregnancy | 18 weeks of pregnancy, 4 weeks post-vaccine, at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Le Doare, MBBS, PhD, Study Chair — St George's, University of London; Manish Sadarangani, MRCPCH, DPHIL, BM.BCh, MA, Study Chair — BC Children's Hospital Research Institute
Locations (1):
- MUJHU Care Ltd, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nakabembe E, Greenland M, Amaral K, Abu-Raya B, Amone A, Andrews N, Cantrell L, Lesne E, Gorringe A, Halkerston R, Mcstraw N, Dixon L, Hunter OF, Heath PT, Imede E, Kyohere M, Musoke P, Nakimuli A, Sekikubo M, Taylor S, Tusubira V, Sadarangani M, Le Doare K. Safety and immunogenicity of an acellular pertussis vaccine containing genetically detoxified pertussis toxin administered to pregnant women living with and without HIV and their newborns (WoMANPOWER): a randomised controlled trial in Uganda. Lancet Glob Health. 2025 Jan;13(1):e81-e97. doi: 10.1016/S2214-109X(24)00409-1. PMID 39706666